CLINICAL TRIAL: NCT05379309
Title: Compliance in Non Invasive Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Karen Funderskov, MScN project nurse, Glostrup University Hospital, Copenhagen
Other Study IDs: COMP1
Record Dates: First submitted 2022-05-11; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Database study of the adherence to treatment to non-invasive mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* patients in non invasive mechanical ventilation and affiliated by the respiratory centre of the East of Denmark
* registered in telemedical solution in the period from 01.01.2020 to 04.01.2022
* Age above 18 years

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Use of treatment more than 4 hr. per day | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Staehr-Rye AK, Irlind TO, Funderskov K, Gatke MR, Kuchen SHL. Adherence to long-term non-invasive positive airway pressure therapy. Dan Med J. 2024 Oct 25;71(11):A04240290. doi: 10.61409/A04240290. PMID 39575944